CLINICAL TRIAL: NCT01822860
Title: The Effect of Chlorthalidone Compared to Hydrochlorothiazide on Endothelial Function in Hypertensive Patients: A Pilot Study
Brief Title: Chlorthalidone Compared to Hydrochlorothiazide on Endothelial Function
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study subjects were not able to be recruited
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-16628
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: Hypertension; Endothelial dysfunction
MeSH Terms: conditions — Hypertension | interventions — Chlorthalidone; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Subjects will receive chlorthalidone, hydrochlorothiazide, and placebo each for 4 weeks in a randomized sequence.
  Interventions: Drug: Placebo
- Chlorthalidone 12.5 mg (Experimental): Subjects will receive chlorthalidone, hydrochlorothiazide, and placebo each for 4 weeks in a randomized sequence.
  Interventions: Drug: Chlorthalidone 12.5 mg
- Hydrochlorothiazide 25 mg (Active Comparator): Subjects will receive chlorthalidone, hydrochlorothiazide, and placebo each for 4 weeks in a randomized sequence.
  Interventions: Drug: Hydrochlorothiazide 25 mg

INTERVENTIONS:
Drug: Chlorthalidone 12.5 mg
  Arms: Chlorthalidone 12.5 mg
Drug: Hydrochlorothiazide 25 mg
  Arms: Hydrochlorothiazide 25 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
Chlorthalidone will result in improved endothelial function compared to hydrochlorothiazide as measured by flow mediated vasodilatation.

DETAILED DESCRIPTION:
This is a randomized, double-blind, crossover study to evaluate chlorthalidone and hydrochlorothiazide and their effects on endothelial function in hypertensive patients. Subjects will receive chlorthalidone 12.5 mg, hydrochlorothiazide 25 mg, and placebo each for 4 weeks with a 1 week washout between study periods. Sequence of study drugs will be randomized. Flow mediated vasodilatation will be measured at baseline and after each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 or older
* Diagnosis of hypertension
* Current blood pressure > 120/80 mm Hg

Exclusion Criteria:

* Use of a thiazide-type diuretic within the last 1 month
* Known allergy to any study medications
* History of gout or hyperuricemia
* SCr >/= 1.8 mg/dl or CrCl < 25 ml/min
* Pregnancy or breastfeeding or planning to become pregnant during study period
* Dementia or cognitive impairment
* Hypokalemia
* Acute coronary syndrome or stroke within 6 months
* Current use of sildenafil, tadalafil, or vardenafil

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Flow mediated vasodilatation | 4 weeks
  Flow mediated vasodilatation will be measured after one month on each drug and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aboeata, MBBCh, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States